CLINICAL TRIAL: NCT02775643
Title: Molecular Analysis of Childhood and Adolescent Melanocytic Lesions
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MACMEL
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: Melanoma; Spitzoid Melanoma; Congenital Melanoma; Melanoma Arising in Giant Nevi; Melanocytic lesions with indeterminate biological behavior; Pigment synthesizing melanomas
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Melanoma tumor tissue and normal blood cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, non-therapeutic study to collect clinical and molecular information of pediatric patients with childhood melanocytic lesions.

PRIMARY OBJECTIVE: To perform a comprehensive molecular analysis of samples either from paraffin embedded and/or frozen tissue from patients with pediatric melanocytic lesions (including melanoma, spitzoid melanoma, congenital melanoma, melanoma arising in giant nevi).

SECONDARY OBJECTIVE: To collect minimal information on patients treated with adjuvant or systemic therapies according to National Comprehensive Cancer Network (NCCN) guidelines.

DETAILED DESCRIPTION:
Investigators will study the DNA and RNA in tumor cells and blood cells to look for changes that may be related to the development of the tumor, as well as changes that may influence how the tumor responds or doesn't respond to treatment. Normal blood cells will be studied to compare to the tumor cells. Investigators will also look at basic information about the treatment received and how the tumor responds, i.e. what kind of chemotherapy, surgery, radiation treatment, or other therapy the participant received, whether they had serious side effects, and how well the tumor responded to the treatment.

As part of regular medical care, tumor will be obtained to determine the type of cancer. For participants who consent to this study, leftover tumor tissue not needed for diagnosis or regular medical care will be studied at St. Jude Children's Research Hospital where scientists will look for changes in the genes of the tumor cells. No additional surgeries or procedures are needed for this study. A small amount of blood (2-3 tablespoons) will be collected and analyzed to determine if the genetic changes in the tumor cells are also found in the blood cells. Small children (<42 lbs.) will have a smaller amount drawn (1-2 tablespoons).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a suspected or confirmed diagnosis of a melanocytic lesion, including:

  * Conventional or "adult-type" melanoma
  * Spitzoid melanoma/atypical Spitz tumor
  * Congenital melanoma
  * Melanoma arising in a giant congenital nevus
  * Melanocytic lesions with indeterminate biological behavior (e.g., pigment synthesizing melanomas)
* Participant was <19 years of age at the time of diagnosis.
* Tissue is available for biologic studies.
* Participant has been enrolled on the TBANK protocol at SJCRH, or will be enrolled before any research tests are performed on their biological materials.

Exclusion Criteria:

* Ocular melanoma
* Inability or unwillingness of research participant or legal guardian to consent.
* Histologic diagnosis other than melanocytic lesion described in 3.1.1.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who meet inclusion criteria and consent to enrollment on the study at St. Jude Children's Research Hospital (SJCRH).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-05-31 (Actual); Primary Completion 2031-05-31 (Estimated); Study Completion 2041-05-31 (Estimated)

PRIMARY OUTCOMES:
Genomic profile | At participant enrollment
  Pathology/molecular samples may be available in pathology banking system or may be obtained at the same time as specimens are taken from individual consenting participants (time varies according to specific therapeutic protocol). A comprehensive molecular analysis of tumor samples either from paraffin embedded and/or frozen tissue from patients will be performed. Summary statistics will be calculated for the pathology/molecular data.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 10 years following on-study date
  OS will be calculated as time from date of diagnosis to date of death or date of last follow-up up to 10 years. OS will be estimated by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pappo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols